CLINICAL TRIAL: NCT05490043
Title: A Phase I Trial of ATG-101 in Patients With Metastatic/Advanced Solid Tumors and Mature B-cell Non-Hodgkin Lymphomas
Brief Title: A Trial of ATG-101 in Patients With Metastatic/Advanced Solid Tumors and Mature B-cell Non-Hodgkin Lymphomas
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The sponsor has decided to adjust the development strategy of the investigational drug in this study.
Sponsor: Antengene (Hangzhou) Biologics Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Antengene Corporation (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATG-101-001-CN
Record Dates: First submitted 2022-07-26; First posted 2022-08-05 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-06

CONDITIONS: Advanced Solid Tumor; Metastatic Solid Tumor; Mature B-cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ATG-101 (Experimental): Dose Escalation Phase:
  Will be conducted with an enhanced PDx cohort.
  Dose Expansion Phase:
  Subjects with advanced or metastatic solid tumors and mature B-NHLs will be enrolled.
  Interventions: Drug: ATG-101

INTERVENTIONS:
Drug: ATG-101 — ATG-101 will be administered intravenously once every 28 days. The dose levels will be determined by the starting dose and the escalation steps taken in the trial. The Dose Expansion Phase will begin at the defined MTD, RP2D, or biologically optimal dose.

SUMMARY:
This is a First-in-Human Phase I trial of ATG-101 in Patients with Metastatic/Advanced Solid Tumors and Mature B-cell Non-Hodgkin Lymphomas.

DETAILED DESCRIPTION:
This is a First-in-Human Phase I trial of ATG-101 in Patients with Metastatic/Advanced Solid Tumors and Mature B-cell Non-Hodgkin Lymphomas. Dose Escalation Phase: Approximately 40-50 subjects with a maximum number of 62; 1-20 subjects for enhanced PDx cohort. Dose Expansion Phase: Estimated between 2 and 5 cohorts, each of approximately 40-50 patients to be expanded.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study-specific procedures, sampling, and analyses.
2. Aged 18 to 75 years as of the date of consent.
3. Histological or cytological confirmation of a solid tumor, and has relapsed or refractory from standard therapies.
4. Subjects with solid tumors have at least 1 measurable lesion per RECIST v1.1.
5. Estimated life expectancy of a minimum of 12 weeks.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 at ICF signature.

Exclusion Criteria:

1. Subjects with CNS tumors or known CNS metastases will be excluded from the Dose Escalation Phase.
2. Prior treatment with a 4-1BB agonist.
3. Subjects with primary liver cancer.
4. Known history of human immunodeficiency virus infection.
5. History of hypersensitivity or history of allergic reactions attributed to drugs with a similar chemical or biologic structure or class to ATG-101.
6. Pregnant or nursing females.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-01-30 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2025-03-17 (Actual)

PRIMARY OUTCOMES:
AEs/SAEs | One year after last patient first dose
  Toxicity will be graded according to the NCI CTCAE, Version 5.0.
DLT (for Dose Escalation Phase only) | One year after last patient first dose
  The DLTs will be evaluated during Cycle 1 of treatment. Toxicity will be graded according to the National Cancer Institute-Common Terminology Criteria for Adverse Events. The DLTs for this study may include the following: Cytokine release syndrome, Hematologic toxicity, Non-hematologic toxicity.

SECONDARY OUTCOMES:
ORR | One year after last patient first dose
  To evaluate preliminary anti tumor activity of ATG-101
DCR | One year after last patient first dose
  To evaluate preliminary anti tumor activity of ATG-101
PFS | One year after last patient first dose
  To evaluate preliminary anti tumor activity of ATG-101
OS | One year after last patient first dose
  To evaluate preliminary anti tumor activity of ATG-101
The incidence of ADA and NAb | One year after last patient first dose
  To evaluate the immunogenicity of ATG-101
Peak Plasma Concentration (Cmax) | One year after last patient first dose
  To evaluate the maximum plasma concentration (Cmax) of ATG-101 in Chinese patient population
Peak Plasma Concentration（Tmax） | One year after last patient first dose
  To evaluate the time to reach Tmax of ATG-101 in Chinese patient population

CONTACTS AND LOCATIONS:
Overall Officials: Hao Cui, MD, Study Director — Medical Physician
Locations (4):
- China (4):
  - Shandong Cancer Hospital, Jinan
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Shanghai Dongfang Hospital, Shanghai
  - Henan Cancer Hospital, Zhengzhou